CLINICAL TRIAL: NCT02849743
Title: Intranasal Oxytocin to Promote Weight Loss in Children, Adolescents, and Adults With Brain Tumors and Hypothalamic Obesity Syndrome
Brief Title: Intranasal Oxytocin in Hypothalamic Obesity
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shana McCormack, MD (Other)
Responsible Party: Sponsor-Investigator, Shana McCormack, MD, Attending Physician, Children's Hospital of Philadelphia
Organization: Children's Hospital of Philadelphia (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 16-012730
Record Dates: First submitted 2016-07-22; First posted 2016-07-29 (Estimated); Results first posted 2022-10-05 (Actual); Last update posted 2022-10-05 (Actual); Status verified 2022-09

CONDITIONS: Craniopharyngioma; Hypothalamic Obesity
Keywords: oxytocin; hypothalamic obesity; craniopharyngioma; metabolism
MeSH Terms: conditions — Craniopharyngioma; Sexual Infantilism | interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Syntocinon (= Oxytocin), then Placebo (Experimental): Week 0 to Week 7: Intranasal oxytocin, administered 3 times per day (at mealtimes) for 8 weeks (dosage based on weight: 16 IU to 24 IU; dose escalation, if appropriate, occurs at 2 weeks)
  Week 8 to Week 11: Washout
  Week 12 to Week 20: Intranasal placebo, administered 3 times per day (at mealtimes) for 8 weeks (dosage based on weight: 16 IU to 24 IU; dose escalation, if appropriate, occurs at 2 weeks)
  *Dose Escalation, as appropriate, at 2 Weeks
  Interventions: Drug: Syntocinon; Drug: Placebo (for Syntocinon)
- Placebo, then Syntocinon (= Oxytocin) (Experimental): Week 0 to Week 7: Intranasal placebo, administered 3 times per day (at mealtimes) for 8 weeks (dosage based on weight: 16 IU to 24 IU; dose escalation, if appropriate, occurs at 2 weeks)
  Week 8 to Week 11: Washout
  Week 12 to Week 20: Intranasal oxytocin, administered 3 times per day (at mealtimes) for 8 weeks (dosage based on weight: 16 IU to 24 IU; dose escalation, if appropriate, occurs at 2 weeks)
  Interventions: Drug: Syntocinon; Drug: Placebo (for Syntocinon)

INTERVENTIONS:
Drug: Syntocinon — The active substance of Syntocinon is a synthetic nonapeptide identical to the posterior pituitary hormone oxytocin.
Drug: Placebo (for Syntocinon) — The placebo is identical to the Syntocinon formulation with the exception of the active compound, i.e., without oxytocin.

SUMMARY:
This research study will test if oxytocin, delivered by nasal spray, will promote weight loss in children, adolescents, and adults with Hypothalamic Obesity as compared to a placebo. The study is divided into two parts. During the first part, subjects will receive either oxytocin or placebo. In the second part, subjects will "cross-over" to receive the other treatment - either oxytocin or placebo. During study visits participants will do blood tests, physical exams, metabolic testing, a MRI scan, and some surveys and questionnaires.

ELIGIBILITY:
Inclusion Criteria:

1. Proficient in English.
2. Males or females age 10 to 35 years, inclusive.
3. Weight ≥ 51 kg.
4. Girls must have a negative urine/serum pregnancy test and post-menarchal girls must use an acceptable method of contraception, including abstinence, a barrier method (diaphragm or condom), Depo-Provera, or an oral contraceptive, for the duration of the study.
5. Hypothalamic obesity, defined for the purposes of this protocol as:

   * previously diagnosed with a brain tumor*
   * currently overweight or obese (BMI > 85%ile for age/sex for < 18 years, BMI > 25 kg/m2 for 18 - 35 years)
   * has at least one other endocrinopathy, indicating hypothalamic damage
   * rate of annualized weight gain during any 6 month period (given variability in clinical course) preceding or after diagnosis and treatment greater than 2 standard deviations above population reference ranges for age and sex.
6. At least 6 months since completion of therapy with stable disease/lack of recurrence.
7. Stable for at least 2 months on any pituitary replacement (e.g., glucocorticoid, thyroid hormone, estrogen/progestin or testosterone, growth hormone, except for adjustments of less than or equal to 20%). (Desmopressin is not required to be stable for 2 months. Participants with DI taking desmopressin are required to have intact thirst and be well-controlled on their current dosing regimen.)
8. Stable for at least 2 months on any appetite-modulating medications (e.g., stimulants).
9. Be able to ambulate independently.
10. Parental/guardian permission (informed consent) and child assent.

Exclusion Criteria:

1. Diabetes insipidus without intact thirst mechanism (i.e., history that participant is not thirsty when hypernatremic and/or continues to be thirsty when hyponatremic, by participant/family and/or practitioner report and medical records) and/or "brittle" diabetes insipidus, defined as requiring >1 admission in the past year and/or any admission within the previous 3 months.
2. Diabetes mellitus requiring insulin or insulin secretagogue. Laboratory values: HgbA1c ≥8%
3. Cardiovascular condition, as defined as any of the following: i) abnormal blood pressure, defined as <3%ile or >97%ile for age, sex and height; ii) history of cardiac arrhythmia or arrhythmia detected on screening ECG; iii) history of heart failure and/or cardiomyopathy; iv) prolonged QTc interval (QTc > 460 msec), and/or long QT syndrome phenotype and/or positive genotype for long QT syndrome pathogenic mutations.
4. Concurrent use of medications known to prolong QTc interval and pose high risk for Torsades de Pointes (TdP) according to the current information available (www.crediblemeds.org). Concomitant medications will be assessed by IDS pharmacist, in collaboration with study cardiologist, if additional clarification is needed. In addition, we require that potential participants be on a stable dose for at least 2 months of any medication with the potential to alter cardiac rhythm to ensure the screening ECG reflects steady-state physiology.
5. History of liver disease, with screening laboratory studies:

   Laboratory values: ALT/SGPT > 3.0X upper limit of normal or AST/SGOT > 3.0X upper limit of normal
6. History of chronic kidney disease, with screening laboratory studies:

   Laboratory values: eGFR < 60 mL/min/1.73m2, as defined by the Schwartz formula
7. Clinically significant anemia, with screening laboratory studies:

   Laboratory values: Hemoglobin < 10 g/dL
8. Seizure in the past 12 months.
9. History of gastrectomy, gastric bypass, small or large bowel resection.
10. History of active substance abuse.
11. Current psychotic disorder and/or suicidality.
12. Supra-physiologic (>15 mg/m2/day) prescribed doses of hydrocortisone equivalent.
13. Anticipated clinical plan to initiate or modify pituitary hormone replacement and/or appetite-modulating drugs during the course of the study.
14. Any investigational drug use within 30 days prior to enrollment.
15. Pregnant or lactating females.
16. Individuals with a known sensitivity to either oxytocin or the components of its formulation.
17. Inability to take an intranasal medication (e.g., recent injury).
18. Parents/guardians or subjects who, in the opinion of the Investigator, may be non-compliant with study schedules or procedures.

Ages: 10 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 18 (Actual)
Dates: Start 2016-10; Primary Completion 2021-04 (Actual); Study Completion 2022-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shana E McCormack, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Once consent was obtained, participants were reviewed for eligibility and inclusion in the trial. Individuals meeting criteria were randomized. In total, 18 participants signed informed consent and completed in-person screening. 5 of 18 were considered ineligible after screening due to: concomitant medications (2), ECG findings (2), and BMI (1).
  Intervention Period 1: Week 0 to Week 7, Washout: Week 8 to Week 11, Intervention Period 2: Week 12 to Week 20.
Groups:
- Syntocinon (= Oxytocin), Then Placebo: 1. Intranasal oxytocin, administered 3 times per day (at mealtimes) for 8 weeks (dosage based on weight: 16 IU to 24 IU; dose escalation, if appropriate, occurs at 2 weeks)
  2. Intranasal placebo, administered 3 times per day (at mealtimes) for 8 weeks (dosage based on weight: 16 IU to 24 IU; dose escalation, if appropriate, occurs at 2 weeks) *Dose Escalation, as appropriate, at 2 Weeks
  Syntocinon: The active substance of Syntocinon is a synthetic nonapeptide identical to the posterior pituitary hormone oxytocin.
  Placebo (for Syntocinon): The placebo is identical to the Syntocinon formulation with the exception of the active compound, i.e., without oxytocin.
- Placebo, Then Syntocinon (= Oxytocin): 1. Intranasal placebo, administered 3 times per day (at mealtimes) for 8 weeks (dosage based on weight: 16 IU to 24 IU; dose escalation, if appropriate, occurs at 2 weeks)
  2. Intranasal oxytocin, administered 3 times per day (at mealtimes) for 8 weeks (dosage based on weight: 16 IU to 24 IU; dose escalation, if appropriate, occurs at 2 weeks)
  Syntocinon: The active substance of Syntocinon is a synthetic nonapeptide identical to the posterior pituitary hormone oxytocin.
  Placebo (for Syntocinon): The placebo is identical to the Syntocinon formulation with the exception of the active compound, i.e., without oxytocin.
Period: First Intervention (8 Weeks)
Arm/Group | Syntocinon (= Oxytocin), Then Placebo | Placebo, Then Syntocinon (= Oxytocin)
Started | 6 | 7
Completed | 6 | 6
Not Completed | 0 | 1
Not completed — Stopping Criteria Met | 0 | 1
Period: Washout (4 Weeks)
Arm/Group | Syntocinon (= Oxytocin), Then Placebo | Placebo, Then Syntocinon (= Oxytocin)
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0
Period: Second Intervention (8 Weeks)
Arm/Group | Syntocinon (= Oxytocin), Then Placebo | Placebo, Then Syntocinon (= Oxytocin)
Started | 6 | 6
Completed | 5 | 6
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Syntocinon (= Oxytocin), Then Placebo | Placebo, Then Syntocinon (= Oxytocin) | Total
Number analyzed (Participants) | 6 | 7 | 13
Age, Continuous [Median (Inter-Quartile Range); unit: Years] | 17.0 [11.9 to 21.4] | 15.3 [14.3 to 16.0] | 15.3 [13.3 to 20.6]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 6
  Male | 4 | 3 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 6 | 5 | 11
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 5 | 6 | 11
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 7 | 13

OUTCOME MEASURES:

1. Primary Outcome: Weight Loss
Description: The primary objective of this study is to determine whether treatment with 8 weeks of intranasal OXT (relative to 8 weeks of placebo) will promote weight loss in children and adolescents with brain tumors and hypothalamic obesity syndrome ages 10 to 35 years. Specifically, the primary outcome will be: the difference of the post-treatment weight between the two periods (treatment vs. placebo); the statistical model will include the difference of the baseline weight between the two periods and the sequence (OXT-PBO versus PBO-OXT).
Time Frame: Assessed at the beginning and end of each Intervention Period (Intervention 1: Visit 1 to Visit 4 = 8 Weeks, Intervention 2: Visit 5 to Visit 8 = 8 Weeks)
Population: In order to be included, participants needed data in Intervention 1 (Block 1) and Intervention 2 (Block 2). 10 of 13 Participants with complete data available for analysis.
Measure: Median (Inter-Quartile Range); unit: kg
Groups:
- Oxytocin: Within Participant Change in Body Weight with Oxytocin for 8 Weeks
- Placebo: Within Participant Change in Body Weight with Placebo for 8 Weeks
Arm/Group | Oxytocin | Placebo
Number analyzed (Participants) | 10 | 10
kg
  Baseline | 88.3 [74.7 to 108.6] | 91.9 [77.9 to 114.6]
  Change at 8 Weeks | 1.2 [0.9 to 1.8] | 0.9 [-0.2 to 1.6]
Statistical Analysis 1: Comparison: Oxytocin vs Placebo; Test type: Other; p = 0.92, Regression, Linear; Least Means Square = -0.5

2. Secondary Outcome: Peripheral Oxytocin Area Under the Curve (AUC)
Description: We will determine the immediate peripheral pharmacokinetics of intranasal oxytocin (versus placebo/endogenous oxytocin). In order to minimize participant burden, each participant had the assessment at one time point with either the low or high dose of oxytocin. And at one point during the placebo block.
  For this exploratory outcome, visits representing lower dose and higher dose oxytocin were Combined versus lower and higher dose placebo.
Time Frame: Assessed during each treatment block: at either initial lower dose at baseline (week 0 & week 12) or increased dose at 2 weeks (week 2 & week 15); 50% of participants at each set.
Population: In order to be included participants had to have samples collected during both Intervention 1 and Intervention 2. IV Access was not able to be obtained in some individuals. 7 of 13 Participants had data available for analysis. Specimens were collected during the lower dose (Visit 1 or Visit 5) or the higher dose (Visit 2 or Visit 6). As this assessment was only administered once per Intervention, we are not able to calculate/report the change at 8 weeks.
Measure: Median (Inter-Quartile Range); unit: Concentration (min*pg/mL)
Groups:
- Oxytocin: Within Participant Difference After Oxytocin in Peripheral Oxytocin (Area Under the Curve)
- Placebo: Within Participant Difference After Placebo in Peripheral Oxytocin (Area Under the Curve)
Arm/Group | Oxytocin | Placebo
Number analyzed (Participants) | 7 | 7
Concentration (min*pg/mL)
  Baseline | 101792 [92722 to 123638] | 99110 [90692 to 132989]
  Change at 8 Weeks | NA [NA to NA] — As this assessment was only administered once per Intervention, we are not able to calculate/report the change at 8 weeks. | NA [NA to NA] — As this assessment was only administered once per Intervention, we are not able to calculate/report the change at 8 weeks.
Statistical Analysis 1: Comparison: Oxytocin vs Placebo; Test type: Other; p = 0.57, Regression, Linear; Regression Coefficient = -15784

3. Other Pre Specified Outcome: Cognitive Restraint at Test Meal Attributable to Oxytocin vs Placebo
Description: Cognitive Restraint at Test Meal Attributable to Oxytocin vs Placebo measured using stop-signal task, stop signal reaction time (SSRT).
  For this exploratory outcome, in order to minimize participant burden, each participant had the assessment at one time point with either the low or high dose of oxytocin. And at one point during the placebo block for comparison.
Time Frame: Intervention 1: Week 2 (Low Dose) or Week 4 (High Dose) and Intervention 2: Week 14 (Low Dose) or Week 16 (High Dose)
Population: In order to be included, participants needed data in Intervention 1 (Block 1) and Intervention 2 (Block 2) in order to be included. 11 of 13 Participants with Data for Analysis. As this assessment was only administered once per Intervention, we are not able to calculate/report the change at 8 weeks.
Measure: Median (Inter-Quartile Range); unit: msec
Groups:
- Oxytocin: Within participant difference in response time (msec) on SSRT with Oxytocin
  Mixed effects model of other outcomes were also constructed. The "treatment duration" variable reflects the time (in days) in within the treatment Block when the outcome was measured.
- Placebo: Within participant difference in response time (msec) on SSRT with Placebo
  Mixed effects model of other outcomes were also constructed. The "treatment duration" variable reflects the time (in days) in within the treatment Block when the outcome was measured.
Arm/Group | Oxytocin | Placebo
Number analyzed (Participants) | 11 | 11
msec
  Baseline | 282 [255 to 326] | 247 [170 to 276]
  Change at 8 Weeks | NA [NA to NA] — SSRT was assessed at either the lower dose (Visit 1 or Visit 5) or the higher dose (Visit 2 or Visit 6). As this assessment was only administered once per Intervention, we are not able to calculate/report the change at 8 weeks. | NA [NA to NA] — SSRT was assessed at either the lower dose (Visit 1 or Visit 5) or the higher dose (Visit 2 or Visit 6). As this assessment was only administered once per Intervention, we are not able to calculate/report the change at 8 weeks.
Statistical Analysis 1: Comparison: Oxytocin vs Placebo; Test type: Other; p = 0.21, Mixed Models Analysis; Regression Coefficient = 48

4. Other Pre Specified Outcome: Within Participant Difference in Calories Consumed Attributable to Oxytocin vs Placebo Dose 1 (Week 0 & Week 12), as a % of kcal Offered.
Description: Within Participant Difference in Calories Consumed Attributable to Oxytocin vs Placebo Dose 1 (Week 0 & Week 12). Total number of calories consumed during the standardized test meal.
Time Frame: Assessed during Intervention 1: Week 0 (Dose 1) and Intervention 2: Week 12 (Dose 1)
Population: In order to be included, participants had to have data in Intervention 1 (Visit 1, Week 0) and Intervention 2 (Visit 5, Week 12). 9 of 13 Participants had data available for analysis. As this assessment was only administered once per Intervention, we are not able to calculate/report the change at 8 weeks.
Measure: Median (Inter-Quartile Range); unit: % of total kcal offered
Groups:
- Oxytocin: Within Participant Difference in Calories Consumed with Oxytocin Dose 1. Total number of kcal eaten, as a % of total kcal offered.
- Placebo: Within Participant Difference in Calories Consumed with Placebo Dose 1. Total number of kcal eaten, as a % of total kcal offered.
Arm/Group | Oxytocin | Placebo
Number analyzed (Participants) | 9 | 9
% of total kcal offered
  Baseline (Week 0 of Intervention) | 72.4 [59.7 to 75.5] | 72.6 [70.9 to 77.7]
  Change at 8 Weeks | NA [NA to NA] — As this assessment was only administered once per Intervention, we are not able to calculate/report the change at 8 weeks. | NA [NA to NA] — As this assessment was only administered once per Intervention, we are not able to calculate/report the change at 8 weeks.
Statistical Analysis 1: Comparison: Oxytocin vs Placebo; Test type: Other; p = 0.55, Regression, Linear; Regression Coefficient = -2.8

5. Other Pre Specified Outcome: Within Participant Difference in Calories Consumed Attributable to Oxytocin vs Placebo Dose 2 (Week 2 & Week 14), as a % of kcal Offered.
Description: Within Participant Difference in Calories Consumed Attributable to Oxytocin vs Placebo Dose 2 (Week 2 & Week 14). Total number of calories consumed during the standardized test meal.
Time Frame: Assessed during Intervention 1: Week 2 (Dose 2) and Intervention 2: Week 14 (Dose 2).
Population: In order to be included, participants had to have data in Intervention 1 (Visit 2, Week 2) and Intervention 2 (Visit 6, Week 14). 9 of 13 Participants had data available for analysis. As this assessment was only administered once per Intervention, we are not able to calculate/report the change at 8 weeks.
Measure: Median (Inter-Quartile Range); unit: % of total kcal offered
Groups:
- Oxytocin: Within Participant Difference in Calories Consumed with Oxytocin Dose 2.
  Total number of kcal eaten, as a % of total kcal offered.
- Placebo: Within Participant Difference in Calories Consumed with Placebo Dose 2.
  Total number of kcal eaten, as a % of total kcal offered.
Arm/Group | Oxytocin | Placebo
Number analyzed (Participants) | 9 | 9
% of total kcal offered
  Week 2 of Intervention | 72.6 [66.3 to 78.3] | 67.7 [55.7 to 78.5]
  Change at 8 Weeks | NA [NA to NA] — As this assessment was only administered once per Intervention, we are not able to calculate/report the change at 8 weeks. | NA [NA to NA] — As this assessment was only administered once per Intervention, we are not able to calculate/report the change at 8 weeks.
Statistical Analysis 1: Comparison: Oxytocin vs Placebo; Test type: Other; p = 0.86, Regression, Linear; Regression Coefficient = 1.2

6. Other Pre Specified Outcome: Within Participant Difference After Oxytocin vs After Placebo in Resting Energy Expenditure (kcal/kg Lean Body Mass/Day)
Description: Within Participant Difference After Oxytocin vs After Placebo in Resting Energy Expenditure (kcal/kg lean body mass/day). Resting Energy Expenditure (REE) with output of kcal/kg lean body mass/day measured using indirect calorimetry.
Time Frame: Assessed at the end of each treatment block: Week 8 & Week 20.
Population: In order to be included, participants had to have data in Intervention 1 (Visit 4, Week 8) and Intervention 2 (Visit 8, Week 20). 9 of 13 Participants had data available for analysis from the end of both treatment blocks.
Measure: Median (Inter-Quartile Range); unit: kcal/kg lean mass/day
Groups:
- Oxytocin: Within Participant Difference After Oxytocin in Resting Energy Expenditure (kcal/kg lean body mass/day) at the end of the Intervention Period (8 Weeks).
  Mixed effects model of other outcomes were also constructed. The "treatment duration" variable reflects the time (in days) in within the treatment Block when the outcome was measured.
- Placebo: Within Participant Difference After Placebo in Resting Energy Expenditure (kcal/kg lean body mass/day) at the end of the Intervention Period (8 Weeks).
  Mixed effects model of other outcomes were also constructed. The "treatment duration" variable reflects the time (in days) in within the treatment Block when the outcome was measured.
Arm/Group | Oxytocin | Placebo
Number analyzed (Participants) | 9 | 9
kcal/kg lean mass/day
  End of Intervention | 129.5 [118.2 to 148.1] | 127.2 [108.3 to 137.9]
  Change at 8 Weeks | NA [NA to NA] — As this assessment was only administered once per Intervention, we are not able to calculate/report the change at 8 weeks. | NA [NA to NA] — As this assessment was only administered once per Intervention, we are not able to calculate/report the change at 8 weeks.
Statistical Analysis 1: Comparison: Oxytocin vs Placebo; Test type: Other; p = 0.88, Regression, Linear; Regression Coefficient = 2.4

7. Other Pre Specified Outcome: Respiratory Quotient (VCO2/VO2)
Description: Within Participant Difference After Oxytocin vs Placebo in Respiratory Quotient (RQ) measured using indirect calorimetry.
Time Frame: Assessed at the end of each treatment block: week 8 & week 20.
Population: In order to be included, participants had to have data in Intervention 1 (Visit 4, Week 8) and Intervention 2 (Visit 8, Week 20). 9 of 13 Participants had data available for analysis from the end of both treatment blocks. SSRT was assessed at either the lower dose (Visit 1 or Visit 5) or the higher dose (Visit 2 or Visit 6). As this assessment was only administered once per Intervention, we are not able to calculate/report the change at 8 weeks.
Measure: Median (Inter-Quartile Range); unit: Ratio (L C02/L 02)
Groups:
- Oxytocin: Within Participant Difference After Oxytocin in Respiratory Quotient (RQ) (VCO2/VO2) at the end of the Intervention (8 Weeks).
- Placebo: Within Participant Difference After Placebo in Respiratory Quotient (RQ) (VCO2/VO2) at the end of the Intervention (8 Weeks).
Arm/Group | Oxytocin | Placebo
Number analyzed (Participants) | 9 | 9
Ratio (L C02/L 02)
  End of Intervention | 0.8 [0.8 to 0.8] | 0.8 [0.8 to 0.9]
  Change at 8 Weeks | NA [NA to NA] — As this assessment was only administered once per Intervention, we are not able to calculate/report the change at 8 weeks. | NA [NA to NA] — As this assessment was only administered once per Intervention, we are not able to calculate/report the change at 8 weeks.
Statistical Analysis 1: Comparison: Oxytocin vs Placebo; Test type: Other; p = 0.50, Regression, Linear; Regression Coefficient = -0.02

8. Other Pre Specified Outcome: Within Participant Difference After Oxytocin vs Placebo in % Body Fat
Description: Total % Body Fat measured using dual energy x-ray absorptiometry (DXA).
Time Frame: Assessed at the end of each treatment block: week 8 & week 20.
Population: In order to be included, participants had to have data in Intervention 1 and Intervention 2. 10 of 13 Participants had data available for analysis. As this assessment was only administered once per Intervention, we are not able to calculate/report the change at 8 weeks.
Measure: Median (Inter-Quartile Range); unit: percent body fat
Groups:
- Oxytocin: Within Participant Difference After Oxytocin in % Body Fat
  Linear regression model.
- Placebo: Within Participant Difference After Placebo in % Body Fat
  Linear regression model.
Arm/Group | Oxytocin | Placebo
Number analyzed (Participants) | 10 | 10
percent body fat
  End of Intervention | 50.1 [44.1 to 54.3] | 50.6 [45.9 to 55.0]
  Change at 8 Weeks | NA [NA to NA] — As this assessment was only administered once per Intervention Period, we are not able to calculate/report the change at 8 weeks. | NA [NA to NA] — As this assessment was only administered once per Intervention Period, we are not able to calculate/report the change at 8 weeks.
Statistical Analysis 1: Comparison: Oxytocin vs Placebo; Test type: Other; p = 0.49, Regression, Linear; Regression Coefficient = -0.02

9. Other Pre Specified Outcome: Skeletal Muscle Oxidative Phosphorylation (OXPHOS) Capacity
Description: Measured using MRI-based post-exercise Creatine Chemical Exchange Saturation Transfer (CrCEST) decline exponential time constant.
Time Frame: Assessed at the end of each treatment block.
Population: Limited data was collected for the skeletal muscle oxidative phosphorylation capacity. The data requires extensive review for quality prior to analysis. The post-processing requirements are extensive. Analyzed data is not available.
Groups:
- Within Participant Change in Skeletal Muscle OXPHOS Capacity Attributable to Oxytocin vs Placebo: Within Participant Change in Skeletal Muscle Oxidative Phosphorylation Capacity Attributable to Oxytocin vs Placebo
Arm/Group | Within Participant Change in Skeletal Muscle OXPHOS Capacity Attributable to Oxytocin vs Placebo
Number analyzed (Participants) | 0

10. Other Pre Specified Outcome: Within Participant Change in Hyperphagia (Total Score) Attributable to Oxytocin vs Placebo
Description: Measured using the Dykens Hyperphagia Questionnaire.
  The Dykens Hyperphagia Questionnaire is a 11-item questionnaire with responses on a scale of 1 to 5. 1 = Not a Problem, 5 = Severe or Frequent Problem. The scale includes three domains: hyperphagic behavior, hyperphagic drive, and hyperphagic severity. There is also a total or overall score which is calculated by combining the scores from each domain. Maximum Possible Score: 55, Minimum Possible Score: 11. Higher scores indicated more severe and/or frequent Hyperphagia.
Time Frame: Assessed using data from Intervention 1: Screening and Visit 4 (Week 8) and Intervention 2: Visit 5 (Week 12) and Visit 8 (Week 20).
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: score on a scale
Groups:
- Oxytocin: Within Participant Change in Hyperphagia (Total Score) with Oxytocin for 8 Weeks.
  Change in overall score on Hyperphagia Questionnaire.
- Placebo: Within Participant Change in Hyperphagia (Total Score) with Placebo for 8 Weeks.
  Change in overall score on Hyperphagia Questionnaire.
Arm/Group | Oxytocin | Placebo
Number analyzed (Participants) | 10 | 10
score on a scale
  Baseline | 20 [15.3 to 27] | 20.5 [16.5 to 23.8]
  Change at 8 Weeks | 2 [-0.8 to 2.8] | 0 [-3.3 to 0.8]
Statistical Analysis 1: Comparison: Oxytocin; Test type: Other; p = 0.68, Regression, Linear; Regression Coefficient = -0.7

11. Other Pre Specified Outcome: Within Participant Change in Disinhibition of Eating Attributable to Oxytocin vs Placebo
Description: Within Participant Change in Disinhibition of Eating Attributable to Oxytocin vs Placebo. Measured using the Eating Inventory questionnaire.
  The Eating Inventory consists of 36 statements where participants respond true or false, 14 questions where participants select a response from 1 (least severe: rarely or not at all) to 4 (most severe: always or very much), one final question askes participants to rate their level of restraint in eating from 1 (no restraint) to 6 (constantly limiting food). The scores are assessed in 3 dimensions: Dietary Restraint (Max Score: 21), Disinhibition (Max Score: 16), and Hunger (Max Score: 14).
  Within Participant Change in Scores from the Disinhibition of Eating dimension are reported.
Time Frame: as for outcome 10
Population: In order to be included, participants needed data in Intervention 1 (Block 1) and Intervention 2 (Block 2). 10 of 13 Participants had complete data available for analysis.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Groups:
- Oxytocin: Within Participant Change in Disinhibition of Eating with Oxytocin for 8 Weeks. Measured using the Eating Inventory.
- Placebo: Within Participant Change in Disinhibition of Eating with Placebo for 8 Weeks. Measured using the Eating Inventory.
Arm/Group | Oxytocin | Placebo
Number analyzed (Participants) | 10 | 10
score on a scale
  Baseline | 8.5 [4.5 to 10.8] | 4 [3.3 to 10.5]
  Change at 8 Weeks | 0 [-1.8 to 0.8] | 0 [-0.8 to 1]
Statistical Analysis 1: Comparison: Oxytocin; Test type: Other; p = 0.52, Regression, Linear; Regression Coefficient = -0.6

12. Other Pre Specified Outcome: Within Participant Change in Mental and Emotional Health Related Quality of Life Attributable to Oxytocin vs Placebo
Description: The National Institute of Neurological Disorders and Stroke (NINDS) quality of life in neurological disorders (Neuro-QoL) scale is a set of self-reported measures to assess health-related quality of life of adults and children.
  Individuals rate domains on a scale from 1 (Never/Not at all) to 5 (Always/Very Often). Each response is assigned a value. Values are combined for a total raw score, then converted to a T-Scores (cohort-specific mean 50, SD 10). Higher scores on the sub-scale domains indicate more of the entity. Adult and child scores were combined in analyses.
Time Frame: as for outcome 10
Population: In order to be included, participants had to have data in Intervention 1 and Intervention 2. 11 of 13 Participants had data available for analysis.
Measure: Median (Inter-Quartile Range); unit: T-Score
Groups:
- Oxytocin: Within Participant Change in Quality of Life Measures with Oxytocin for 8 Weeks. Measured using the Neuro-QoL scale.
- Placebo: Within Participant Change in Quality of Life Measures with Placebo for 8 Weeks. Measured using the Neuro-QoL scale.
Arm/Group | Oxytocin | Placebo
Number analyzed (Participants) | 11 | 11
T-Score
  Baseline: Anxiety | 49.9 [47.7 to 52.8] | 45.7 [37.5 to 55.6]
  Change at 8 Weeks: Anxiety | -2 [-4.6 to 0.7] | 0 [0 to 0]
  Baseline: Depression | 42 [36.4 to 49.7] | 36.4 [36.4 to 49.9]
  Change at 8 Weeks: Depression | 0 [0 to 3.1] | 0 [0 to 1.2]
  Baseline: Cognition | 50.4 [48.6 to 56.6] | 44 [39.8 to 51.7]
  Change at 8 Weeks: Cognition | 0 [-4.1 to 0] | 1.2 [0 to 2]
  Baseline: Social Function (Adults) or Peer Interaction (Children) | 47.9 [45.1 to 51.4] | 47.9 [38.6 to 60.2]
  Change at 8 Weeks: Social Function | -1.6 [-4.9 to 0] | -1.8 [-9.6 to 0]
Statistical Analysis 1: Comparison: Oxytocin; Neuro-QoL - Anxiety; Test type: Other; p = 0.91, Regression, Linear; Regression Coefficient = -0.2
Statistical Analysis 2: Comparison: Oxytocin; Neuro-QoL - Depression; Test type: Other; p = 0.91, Regression, Linear; Regression Coefficient = -0.2
Statistical Analysis 3: Comparison: Oxytocin; Neuro-QoL - Cognition; Test type: Other; p = 0.04, Regression, Linear; Regression Coefficient = 4.7
Statistical Analysis 4: Comparison: Oxytocin; Neuro-QoL - Social Function; Test type: Other; p = 0.36, Regression, Linear; Regression Coefficient = 2.3

13. Other Pre Specified Outcome: Within Participant Change in Family Assessment Device-General Function Scale (FAD-GFS) Attributable to Oxytocin vs Placebo
Description: Within Participant Change in Family Assessment Device-General Function Scale (FAD-GFS) Attributable to Oxytocin vs Placebo.
  The Family Assessment Device (FAD-GFS) includes 12 statements where individuals select from a scale of 4 responses ranging from Strongly Agree (SA) to Strongly Disagree (SD). Each response has a score ranging from 1 to 4, some of the items are reverse scored (i.e. 1 = 4, 2 = 3, 3 = 2, 4 = 1). Minimum Total Score: 12, Maximum Total Score: 48. The scores for each question are added and then divided by the total number of questions. The Minimum Overall Score: 1, Maximum Overall Score: 4. A score of 2 or above is considered dysfunction.
Time Frame: as for outcome 10
Population: In order to be included, participants had to have data in Intervention 1 and Intervention 2. 9 of 13 Participants had data available for analysis. This assessment was administered for participants who lived in the same house as the caregiver who would complete the assessment.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Groups:
- Oxytocin: Within Participant Change in Family Assessment Device-General Function Scale (FAD-GRS) with Oxytocin for 8 Weeks
- Placebo: Within Participant Change in Family Assessment Device-General Function Scale (FAD-GRS) with Placebo for 8 Weeks
Arm/Group | Oxytocin | Placebo
Number analyzed (Participants) | 9 | 9
score on a scale
  Baseline | 1.6 [1 to 2.3] | 1.4 [1.1 to 1.8]
  Change at 8 Weeks | -0.1 [-0.5 to 0.1] | 0 [0 to 0.2]
Statistical Analysis 1: Comparison: Oxytocin; Test type: Other; p = 0.64, Regression, Linear; Regression Coefficient = 0.05

14. Other Pre Specified Outcome: Within Participant Change in Voluntary Physical Activity Attributable to Oxytocin vs Placebo
Description: Measured using the Bone Mineral Density in Childhood Study (BMDCS) physical activity questionnaire.
  The Bone Mineral Density in Childhood Study (BMDCS) questionnaire captures the amount of time spent in physical activity. The assessment asks participants to record the number of hours spent in different categories of physical activity (Min: 0 hours per week, Max: 11+ hours per week).
Time Frame: as for outcome 10
Population: In order to be included, participants had to have data in Intervention 1 and Intervention 2. 10 of 13 Participants had data available for analysis.
Measure: Median (Inter-Quartile Range); unit: hours per week of physical activity
Groups:
- Oxytocin: Median change reported in physical activity, time spent in any activity (hours per week), with Oxytocin.
- Placebo: Median change reported in physical activity, time spent in any activity (hours per week), with Placebo.
Arm/Group | Oxytocin | Placebo
Number analyzed (Participants) | 10 | 10
hours per week of physical activity
  Baseline | 1.3 [1.2 to 2] | 1.1 [0.3 to 1.5]
  Change at 8 Weeks | -0.4 [-1.6 to -0.08] | -0.1 [-0.6 to 0.3]
Statistical Analysis 1: Comparison: Oxytocin; Test type: Other; p = 0.83, Regression, Linear; Regression Coefficient = 0.05

15. Other Pre Specified Outcome: Eye-Tracking Task
Description: Amount of time spent viewing socially relevant versus socially irrelevant stimuli during eye-tracking.
Time Frame: Assessed at the end of each treatment block.
Population: Limited data was collected for the Eye Tracking Task. The data requires extensive review for quality prior to analysis. The post-processing requirements are extensive. Analyzed data is not available.
Groups:
- Within Participant Change in Eye Tracking Attributable to Oxytocin vs Placebo: Within Participant Change in Eye Tracking Attributable to Oxytocin vs Placebo
Arm/Group | Within Participant Change in Eye Tracking Attributable to Oxytocin vs Placebo
Number analyzed (Participants) | 0

16. Other Pre Specified Outcome: EEG Task
Description: N170 EEG signal during eye-tracking
Time Frame: Assessed at the end of each treatment block.
Population: EEG task was not completed due to difficulties with equipment. No data collected for analysis.
Arm/Group | Syntocinon (= Oxytocin), Then Placebo | Placebo, Then Syntocinon (= Oxytocin)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse Event data were collected from the time of informed consent through the duration of participation (Up to 20 Weeks).
Description: The Safety Monitoring Uniform Report Form (SMURF) was administered at each in-person visit and each telephone check-in visit to assess OXT specific side effects. The full SMURF contains a general inquiry, several questions about daily activities, and modified questions specific to potential OXT side effects.
Groups:
- Syntocinon (Intranasal Oxytocin): 1) Intranasal oxytocin, administered 3 times per day (at mealtimes) for 8 weeks (dosage based on weight: 16 IU to 24 IU; dose escalation, if appropriate, occurs at 2 weeks)
  Syntocinon: The active substance of Syntocinon is a synthetic nonapeptide identical to the posterior pituitary hormone oxytocin.
- Placebo: 1) Intranasal placebo, administered 3 times per day (at mealtimes) for 8 weeks (dosage based on weight: 16 IU to 24 IU; dose escalation, if appropriate, occurs at 2 weeks)
  Placebo (for Syntocinon): The placebo is identical to the Syntocinon formulation with the exception of the active compound, i.e., without oxytocin.
- Overall: All Participants from Both Treatment Groups.
Arm/Group | Syntocinon (Intranasal Oxytocin) | Placebo | Overall
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 12/12 | 12/12 | 12/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Syntocinon (Intranasal Oxytocin) (N=12) | Placebo (N=12) | Overall (N=12)
Fatigue (General disorders) | 2 (2) | 0 (0) | 2 (2)
Irritability (Psychiatric disorders) | 1 (1) | 1 (1) | 2 (2)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 3 (3) | 3 (3)
Rectal Irritation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Worsening Irritable Bowel Syndrome (IBS) (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Electrocardiogram QT Corrected Interval Prolonged (Cardiac disorders) | 2 (2) | 3 (3) | 5 (5)
Allergic Rhinitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 2 (2)
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 4 (4)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1) | 2 (2)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Dry Lips (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Eye Disorders - Other (Possible Disc Blurring, Eyelid Twitching) (Eye disorders) | 2 (2) | 0 (0) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 2 (2)
Infections - Other (Pharyngitis, Sinusitis) (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Investigations - Other (Low Free T4) (Investigations) | 1 (1) | 2 (2) | 3 (3)
Investigations - Other (Elevated AST) (Investigations) | 1 (1) | 0 (0) | 1 (1)
Investigations - Other (Elevated Bilirubin) (Investigations) | 0 (0) | 1 (1) | 1 (1)

LIMITATIONS AND CAVEATS:
A new package insert for intranasal oxytocin was released indicating a possible risk for QTc prolongation when administered with other medications known to prolong the QTc. In response with advise from our study cardiologist, we revised exclusion criteria, and added post-dose ECG studies to monitor acute effects. These activities impacted recruitment, as did the COVID-19 pandemic, thus target sample size is less than originally planned (see statistical plan for details).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2019-08-20): https://cdn.clinicaltrials.gov/large-docs/43/NCT02849743/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-30): https://cdn.clinicaltrials.gov/large-docs/43/NCT02849743/SAP_001.pdf
  • Informed Consent Form (2020-10-21): https://cdn.clinicaltrials.gov/large-docs/43/NCT02849743/ICF_002.pdf